CLINICAL TRIAL: NCT01456377
Title: A Prospective Controlled Study Randomized Double Blind Study, Evaluate the Effectiveness of Oral Corticosteroids in the Treatment of Stenosis of Lumbar Canal In Symptomatic Patients
Brief Title: The Effectiveness of Oral Corticosteroids in the Treatment of Lumbar Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Luiz Claudio Lacerda Rodrigues, assisten os spine surgeon group, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1892/10
Record Dates: First submitted 2011-10-12; First posted 2011-10-20 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2011-10

CONDITIONS: Spinal Stenosis of Lumbar Region
Keywords: lumbar stenosis; systemic corticosteroids; outcome; security
MeSH Terms: conditions — Constriction, Pathologic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- corticosteroids, analgesics oral pill (Active Comparator): Oral Corticosteroids and oral analgesics
  Interventions: Drug: predinose oral
- placebo (Placebo Comparator): oral placebo and oral analgesics
  Interventions: Drug: placebo group

INTERVENTIONS:
Drug: predinose oral — 1 mg for kg for 3 wekees
  Arms: corticosteroids, analgesics oral pill
Drug: placebo group — use a oral placebo
  Arms: placebo

SUMMARY:
The aim of this study is to evaluate the effectiveness of the use of systemic corticosteroids administered orally in narrow lumbar canal syndrome.

DETAILED DESCRIPTION:
60 patients are being randomized, plank by randomization, the patient and the examiner will be blinded. Will be placed in opaque brown envelopes in order to maintain the secrecy of allocation.

Included patients aged between 50 and 75 years of both sexes participate in the work to accept and sign the Informed Consent The patient will be screened in advance after the acceptance of it will be an anthropometric assessment, with assessment of height, weight and presence of associated comorbidities.

After clinical evaluation they headed for the initial evaluation, after this evaluation, patients are randomized and and delivered to the patient the medication with corticosteroids or placebo for an unrelated medical research. It is also given a bottle of paracetamol 750 mg and a sheet dated, in which the patient is instructed to register the day this sheet and number of capsules taken, which is also an evaluation factor.

evaluation VAS SF 36 Roland Morris questionnaire Test 6-minute walk Likert scale ELegibility Criteria

Clinical diagnosis:

Low back pain and at least two of the following complaints in lower limbs: pain, weakness, burning or numbness that worsens with walking and improves with the cessation of walking.

Radiological diagnosis:

Presence of lumbar canal stenosis with an area less than 100mm2 Hamanishi based on criteria measured at lumbar spine MRI in the follow-up from L1 to S1.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain and at least two of the following complaints in lower limbs: pain, weakness, burning or numbness that worsens with walking and improves with the cessation of walking.

Exclusion Criteria:

* decompensated diabetes mellitus.
* Systemic hypertension and decompensated heart
* systemic disease affecting the lower limbs
* Neuromuscular Disease
* Use of steroids in the past 3 months.
* Patients with previous surgery of the thoracic or lumbar spine.
* cognitive disorder that interferes with the ability to understand or interpret the questionnaires
* Spondylolisthesis except degenerative
* degenerative scoliosis with Cobb angle of 10 °

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-02 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
effectiveness of oral corticosteroids in the treatment of spinal stenosis | 3 months
  The aim of this study is to evaluate the effectiveness of the use of systemic corticosteroids administered orally in narrow lumbar stenosis.
  use SF-36 VAS roland Moris questionnaire

SECONDARY OUTCOMES:
effectiveness and security of oral corticosteroids in the treatment of spinal stenosis | 3 months
  assess the safety of oral corticosteroids in patients with spinal stenosis and tolerability of patients with this medication control of sistemic diseases and safety with oral corticosteroids evaluation for osteoporotic patients in use of oral costicosteroids SF-36 VAS Roland Moris questionnaire 6 minuts walk test

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Santa Marcelina Hospital, São Paulo, São Paulo
  - Santa Mareclina Hospital, São Paulo, São Paulo